CLINICAL TRIAL: NCT06327022
Title: Effects of Social Media-based Electronic Bibliotherapy on Improving the Well-being of Informal Caregivers of People With Dementia
Brief Title: Social Media-based Electronic Bibliotherapy for Dementia Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: P0038444
Record Dates: First submitted 2024-02-18; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-02

CONDITIONS: Mental Health; Quality of Life; Dementia Caregivers
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social media-based electronic bibliotherapy (Experimental): Eight weekly sessions of social media-based electronic bibliotherapy
  Interventions: Other: Social media-based electronic bibliotherapy
- Usual care (Other): Routine services provided by community centers
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Social media-based electronic bibliotherapy — Eight weekly sessions of bibliotherapy are delivered via their daily social media.
  Arms: Social media-based electronic bibliotherapy
Other: Usual care — The routine services provided by community centers
  Arms: Usual care

SUMMARY:
This study aims to assess the efficacy of social media-based electronic bibliotherapy in improving the well-being of informal caregivers of people with dementia compared to a control group.

DETAILED DESCRIPTION:
This randomized controlled trial aims to assess the efficacy of social media-based electronic bibliotherapy in improving the well-being of informal caregivers. Sixty informal caregivers of people with dementia were recruited and randomly allocated to the social media-based electronic bibliotherapy group or usual care group. Participants in the social media-based electronic bibliotherapy group received eight weekly e-bibliotherapy sessions. The control group only accepted the usual care provided by community services, but they received the same intervention materials as the intervention group after project completion. Mental health, caregiving appraisal, health-related quality of life, and psychological well-being were measured to test the intervention's effects immediately after completion. Individual interviews were conducted to explore caregivers' experiences participating in this study within two weeks after completing the intervention.

ELIGIBILITY:
Inclusion Criteria:

* caregivers providing regular care to individuals with mild to moderately severe dementia (Global Deterioration Scale=4~6 of any type), requiring at least five hours per week for a minimum duration of six months;
* aged 18 or above;
* not receiving payment for caregiving services rendered;
* assisting with at least one daily activity of the care recipient;
* possessing reading ability;
* utilized social media platforms such as WhatsApp, Facebook, Twitter, Instagram, and WeChat for over six months.

Exclusion Criteria:

* caregivers with unstable physical or mental conditions;
* caregivers unable to communicate logically;
* involvement in another interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in mental health | Pre-intervention, post-intervention (i.e., within one week after completing the intervention)
  Mental health will be measured with the Depression Anxiety Stress Scale-21. It is a 4-point Likert scale consisting of 21 items that measure levels ofdepression, anxiety, and stress in participants. Higher scores indicategreater severity of mental health problems.

SECONDARY OUTCOMES:
Changes in health related quality of life | Pre-intervention, post-intervention (i.e., within one week after completing the intervention)
  The health-related quality of life will be assessed using the 12-item Short Form Survey. It comprises two domains, namely the physical component summary and the mental component summary. Higher scores indicate better health-related quality of life.
Changes in caregiving appraisal | Pre-intervention, post-intervention (i.e., within one week after completing the intervention)
  Caregiving appraisal will be assessed using the Caregiving Appraisal Scale. It is a 26-item Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Higher scores on this scale indicate more positive caregiving appraisal.
Changes in psychological wellbeing | Pre-intervention, post-intervention (i.e., within one week after completing the intervention)
  The psychological well-being will be assessed using the shorter Chinese version of Ryff's psychological well-being scale. This scale is a Likert 6-point scale (1=strongly disagree, 6=strongly agree) comprising 18 items. Higher scores indicate greater levels of psychological well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Shanshan, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang S, Cheung DSK, Leung SHI, Fan AYN, Ning W, Leung AYM. Social media-based bibliotherapy for improving the mental health of informal caregivers of people with dementia: a randomized controlled trial. BMC Nurs. 2025 Apr 9;24(1):396. doi: 10.1186/s12912-025-02778-7. PMID 40205579